## Official Title of Study:

PH III Study of Lenalidomide and Dexamethasone With or Without Elotuzumab to Treat Previously Untreated Multiple Myeloma (ELO 1 Substudy)

NCT Number: NCT01891643

Document Date (Date in which document was last revised): February 19, 2013



## 6 STATISTICAL ANALYSIS

CS1 level on the cell surface is measured by mean fluorescent intensity.

The level of CS1 protein expression on the surface of bone marrow-myeloma cells and peripheral blood myeloma cells at baseline and at progression, and the change in CS1 level, from baseline to progression, will be summarized, by arm, via descriptive statistics, including the mean, standard deviation, median, inter-quartile range, minimum and maximum. The level of CS1 on the surface of bone marrow-derived myeloma cells and circulating myeloma cells at progression will be regressed on treatment, baseline CS1 level, and treatment by baseline CS1 level interaction to determine whether treatment affects CS1 level at progression, and, if so, whether the magnitude of the effect differs by baseline CS1 level. More complex modeling techniques may be employed, if necessary, such as adding higher order terms for baseline CS1 expression or doing regression on log-transformed CS1 expression.

